CLINICAL TRIAL: NCT01386177
Title: Interactive Effects of Doxazosin and 3,4-Methylenedioxymethamphetamine (MDMA) in Healthy Subjects
Brief Title: Pharmacological Interaction Between Doxazosin and Methylenedioxymethamphetamine (MDMA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 65/11
Record Dates: First submitted 2011-06-03; First posted 2011-06-30 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Mood Disorder; Substance-Related Disorders; Amphetamine-Related Disorders
Keywords: MDMA; doxazosin; norepinephrine; alpha1- receptor; ecstasy; stimulants
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- doxazosin, MDMA, placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: Doxazosin; Drug: placebo

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — 125 mg per os, single dose
  Other Names: MDMA; ecstasy
Drug: Doxazosin — 3 days (-64h) before MDMA: 4 mg doxazosin per os. 2 days (-40h) before MDMA: 8 mg doxazosin per os.
  1 day (-16h) before MDMA: 8 mg doxazosin per os.
  Other Names: Cardura
Drug: placebo — capsules identical to MDMA or doxazosin

SUMMARY:
The purpose of this study is to determinate the effect of a pre-treatment with doxazosin, a alpha1-adrenergic receptor blocker, on the pharmacodynamics and pharmacokinetics of 3,4-methylenedioxymethamphetamine (MDMA, "ecstasy"). The investigators hypothesize that doxazosin will attenuate the cardiovascular and subjective response to MDMA.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is widely used by young people for its euphoric effects. MDMA releases serotonin (5-HT), dopamine, and norepinephrine (NE). NE release is thought to mediate the cardiovascular effects of MDMA and may also contribute to its psychostimulant effects. However, the functional role of adrenergic postsynaptic receptors in the cardiovascular and subjective effects of MDMA in humans is largely unclear. To determine the role of alpha-adrenergic receptors in the response to MDMA in humans the investigators test the effects of the alpha1-receptor blocker doxazosin on the physiological and subjective effects of MDMA. The investigators use a randomized double-blind placebo-controlled cross-over design with four experimental sessions. doxazosin or placebo will be administered before MDMA or placebo to 16 healthy volunteers. Subjective and cardiovascular responses will be repeatedly assessed throughout the experiments and plasma samples are collected for pharmacokinetics. The primary hypothesis is that doxazosin will significantly reduce the blood pressure response to MDMA.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except Tetrahydrocannabinol-containing products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure (mmHg) during 6 hours | 6 hours

SECONDARY OUTCOMES:
Subjective effects during 6 hours | 6 hours
  subjective effects are going to be assessed by various standardized questionnaires (e.g. visual analogue scales (VAS), the 5 dimension Altered State of consciousness questionnaire, or the adjective mood rating scale (AMRS).)
Neuroendocrine plasma levels during 6 hours | 6 hours
  neuroendocrine parameters assessed: prolactin, cortisol, epinephrine, norepinephrine, oxytocin, pro-vasopressin, vasopressin, estrogen,and progesterone
MDMA plasma levels during 6 hours | 6 hours
Genetic polymorphisms | assessed after study completion
  Effects of MDMA on genetic polymorphisms
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

OTHER OUTCOMES:
Prosocial behavior | 5 hours
  Effects on prosociality will be assessed by the Social Value Orientation slide-measurement test.
Empathy | 5 hours
  Emotional empathy will be assessed by the Multifaceted Empathy Test (MET). Cognitive empathy will be assessed by Facial Emotion Recognition Tests and the MET.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Hysek CM, Fink AE, Simmler LD, Donzelli M, Grouzmann E, Liechti ME. alpha(1)-Adrenergic receptors contribute to the acute effects of 3,4-methylenedioxymethamphetamine in humans. J Clin Psychopharmacol. 2013 Oct;33(5):658-66. doi: 10.1097/JCP.0b013e3182979d32. PMID 23857311
- [Derived] Hysek CM, Liechti ME. Effects of MDMA alone and after pretreatment with reboxetine, duloxetine, clonidine, carvedilol, and doxazosin on pupillary light reflex. Psychopharmacology (Berl). 2012 Dec;224(3):363-76. doi: 10.1007/s00213-012-2761-6. Epub 2012 Jun 15. PMID 22700038